CLINICAL TRIAL: NCT05110612
Title: Episodic Future Thinking Intervention Targeting Loss Aversion and Cigarette Smoking
Brief Title: Episodic Future Thinking, Loss Aversion and Cigarette Smoking
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Eric A Thrailkill, Research Assistant Professor, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: FP00002058
Record Dates: First submitted 2021-10-20; First posted 2021-11-08 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Tobacco Smoking
MeSH Terms: conditions — Tobacco Smoking

STUDY DESIGN:
Intervention Model Description: Randomized parallel group design
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Extended Episodic Future Thinking (Experimental): Participants will receive Episodic Future Thinking practice for 8 sessions.
  Interventions: Behavioral: Episodic Future Thinking
- Brief Episodic Future Thinking (Experimental): Participants will receive Episodic Future Thinking practice for 2 sessions.
  Interventions: Behavioral: Episodic Future Thinking
- Control (Sham Comparator): Participants will receive sham Episodic Recent Thinking intervention.
  Interventions: Behavioral: Control Episodic Thinking

INTERVENTIONS:
Behavioral: Episodic Future Thinking — Episodic Future Thinking involves generating positive, autobiographical events that could realistically occur following each of five delays in the subsequent DD task: 1 day, 1 week, 1 month, 3 months, and 1 year. Participants will be told to not include events related specifically to smoking. Using a five-point Likert scale, participants will rate each event according to four dimensions: vividness, enjoyment, importance, and excitement. The event rated the most vivid at each time frame will be chosen for use in subsequent behavioral testing (ties will be settled randomly). Participants will then be recorded reciting a self-created two or three-sentence summary of each event. These recordings will serve as audio cues. Participants will also create abbreviated versions of each description to serve as text cues.
  Arms: Brief Episodic Future Thinking; Extended Episodic Future Thinking
Behavioral: Control Episodic Thinking — Control Episodic Thinking will report three real, positive events that occurred earlier in the session while playing mobile video games. Participants will be told to not include events related specifically to smoking. Using a five-point Likert scale, participants will rate each event according to four dimensions: vividness, enjoyment, importance, and excitement. The event rated the most vivid at each time frame will be chosen for use in subsequent behavioral testing (ties will be settled randomly). Participants will then be recorded reciting a self-created two or three-sentence summary of each event. These recordings will serve as audio cues. Participants will also create abbreviated versions of each description to serve as text cues.
  Arms: Control

SUMMARY:
Controlled laboratory experiment to examine whether Episodic Future Thinking influences loss aversion and cigarette smoking among adult individuals who currently smoke cigarettes daily.

DETAILED DESCRIPTION:
Specific Aim 1: Examine in a controlled laboratory study using a randomized parallel-group design whether an intervention that increases LA among 138 current adult daily cigarette smokers (≥21 years; 50% male/50% female) also (1) decreases cigarette smoking and (2) can improve with practice and (3) sustain effectiveness at a follow-up assessment. Potential influence of DD, other self-control, and potential sociodemographic confounders will be accounted for in all analyses.

Hypothesis 1.1: EFT will increase LA and reduce cigarette smoking (i.e., smoking rate). (Primary) Hypothesis 1.2: Changes in LA will mediate the effect of EFT on cigarette smoking independent of changes in DD, and relevant self-control related factors. (Primary) Hypothesis 1.3: EFT effects will be greater following Extended compared to Brief training. (Secondary) Hypothesis 1.4: Changes in LA and smoking rate sustained at follow up will be mediated by EFT habit learning indexed by the perceived automaticity of cue generation with extended EFT practice. (Exploratory)

ELIGIBILITY:
Inclusion/Exclusion Criteria

Inclusion criteria:

1. Adult ≥ age 21 years.
2. Able to provide informed, written consent.
3. Smoke an average of at least five (5) cigarettes per day for at least one year.
4. Breath CO levels > 8 ppm. If breath CO is less than 8 ppm, we will administer a urine test (NicAlert Strip) and include if result is greater than 2.
5. Desire to quit smoking, but not actively trying to quit or currently taking medications to aid smoking cessation (e.g, varenicline, bupropion).
6. US citizen or a permanent resident alien with a green card
7. Comfortable reading and writing in English

Exclusion criteria:

1. Currently seeking treatment for smoking cessation.
2. Use of tobacco products other than traditional combusted cigarettes on more than 9 of the previous 30 days
3. Positive urine toxicological screen for illicit drug use (i.e., amphetamine, methamphetamine, cocaine, barbiturates, benzodiazepines, buprenorphine, opiates, methadone, oxycodone, phencyclidine).

a. A positive test for marijuana (THC) will not result in exclusion from the study.

d) Breath alcohol level (BAL) at <.01 (Alco-Sensor IV, Intoximeter, Inc., St Louis, MO) at intake.

a. Participants failing the toxicological screen will be allowed to re-screened for the study. These participants will complete the informed consent process an additional time before being re-screened.

e) Recent or current psychiatric episode to be determined with DSM-V criteria. f) Non-correctable vision or hearing impairments. g) Inability to independently read and comprehend written materials (consent form, other study materials and measures).

h) Currently pregnant (to be determined with a pregnancy test) or trying to become pregnant.

i) Currently breastfeeding. j) Exclusive use of "roll your own" cigarettes.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Loss aversion | 30 days
  Loss aversion will be measured with a gamble task developed by Tom et al. (2007). Participants will choose whether to accept or reject each of a series of hypothetical lotteries offering a 50-50 chance of a monetary loss and a monetary gain. Participants will indicate their decision to play a lottery by clicking on accept or reject buttons (strongly accept, accept, reject, strongly reject) located on the screen below the amounts (Figure 2). The task will consist of a series of 49 trials presenting each combination of 7 possible gains (+$2, +$12, +$22, +$32, +$42, +$52, and +$62) and 7 possible losses (-$1, -$6, -$11, -$16, -$21, -$26, and -$31). Combinations of gains and losses will be presented in random order.
Cigarette self-administration | 30 days
  All participants will complete a 60-min self-administration task, in which they can earn single cigarette puffs for every 10 clicks on a moving circle on a computer screen. After completing each response requirement, participants will self-administer 1 cigarette puff. Target cigarette puff volume will be standardized at approximately 70 mL and participants will be instructed to light a cigarette without inhaling, place it in a cigarette holder connected to the pressure sensor, and inhale from the cigarette while estimated puff volume is displayed on the computer screen in real time. The displayed puff volume will turn from white to red at 60 ml and signal the approximate time participants should stop inhaling to reach 70 ml. Participants will have practiced this procedure prior to the task. Participants will be instructed that they can smoke as much or as little as they want during the task.

SECONDARY OUTCOMES:
Delay discounting | 30 days
  Delay discounting will be measured with a standard adjusting-amount task. This task used to measure intervention effects on delay discounting (e.g., Stein et al., 2016). At each of five delays, participants will choose between two different hypothetical amounts: $1,000.00 available after a delay or a smaller amount of money available immediately. The smaller amount will be titrated across six consecutive trials until reaching a point of subjective equality between choice options. Delays will be presented in random order. The value of the smaller amount at indifference indexes the discounted value of the larger option at each delay. This titration process will repeat at each of five delays: 1 day, 1 week, 1 month, 3 months, and 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: ERIC A THRAILKILL, PHD, Principal Investigator — University of Vermont

IPD SHARING:
Plan to Share IPD: Yes
During the study period data will be accessible only to University of Vermont Institutional Review Board-approved research personnel. After all participants complete the study, all data are collected, and the primary results have been published, de-identified data will be made available to other qualified investigators upon request and in a Open Science Foundation repository. Each request will be reviewed and evaluated individually by the PI to ensure that it meets reasonable demands of scientific integrity.
Supporting Information: Study Protocol
Time Frame: Materials will be made available on a perpetual OSF repository after notice of publication.
Access Criteria: Open access

REFERENCES:
- [Background] Stein JS, Wilson AG, Koffarnus MN, Daniel TO, Epstein LH, Bickel WK. Unstuck in time: episodic future thinking reduces delay discounting and cigarette smoking. Psychopharmacology (Berl). 2016 Oct;233(21-22):3771-3778. doi: 10.1007/s00213-016-4410-y. Epub 2016 Aug 23. PMID 27553824
- [Background] Tom SM, Fox CR, Trepel C, Poldrack RA. The neural basis of loss aversion in decision-making under risk. Science. 2007 Jan 26;315(5811):515-8. doi: 10.1126/science.1134239. PMID 17255512